CLINICAL TRIAL: NCT05679765
Title: Analgesic Efficacy of Ultrasound-guided Greater Occipital Nerve Block in Patients of Chronic Migraine
Brief Title: Efficacy of GONB in Patients of Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pain Medicine Department (Other)
Responsible Party: Principal Investigator, Moazzam Ali, Doctor, Head Of Department, Pain Medicine Department
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GONB for migraine
Record Dates: First submitted 2022-12-07; First posted 2023-01-11 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Chronic Migraine; Headache
MeSH Terms: conditions — Headache | interventions — Dexamethasone; Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group G (Experimental): Greater occipital nerve block (GONB) under ultrasound guidance with lidocaine and dexamethasone on the side of headache
  Interventions: Drug: Greater Occipital Nerve Block with dexamethasone and lidocaine; Drug: Greater Occipital Nerve Block with 0.9% saline
- Group S (Active Comparator): Greater occipital nerve block (GONB) under ultrasound guidance on the side of headache with 0.9% Saline (Placebo)
  Interventions: Drug: Greater Occipital Nerve Block with dexamethasone and lidocaine; Drug: Greater Occipital Nerve Block with 0.9% saline

INTERVENTIONS:
Drug: Greater Occipital Nerve Block with dexamethasone and lidocaine — Ultrasound guided Greater occipital nerve block on the side of headache
  Other Names: GONB with dexamethasone and lidocaine
Drug: Greater Occipital Nerve Block with 0.9% saline — Ultrasound guided Greater occipital nerve block on the side of headache
  Other Names: GONB with 0.9% saline

SUMMARY:
The study was carried to determine the analgesic efficacy of greater occipital nerve block in patients of migraine. It was a randomised controlled which took place from april 2022 - october 2022. Fifty patients suffering from migraine were included in the study. Patients in Group G were given greater occipital nerve block (GONB) with lignocaine and dexamethasone under ultrasound guidance while those in Group S were given saline 0.9% as placebo. Pain score using Numeric Rating Scale and number of headache days was assessed at four,eight and twelve weeks after the procedure as a primary outcome. Total headache days were recorded as a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 to 60 years
* diagnosed case of migraine

Exclusion Criteria:

* Patients with known allergies to local anaesthetics
* pregnancy
* history of cranial or cervical surgery
* head injury
* headaches secondary to medication overuse
* patients with uncontrolled systemic disease like blood pressure, diabetes mellitus
* hypo or hyperthyroidism
* patient who had already received GONB or botulinum toxin type A therapy within last 6 months
* major psychiatric disorder
* history of chronic pain syndromes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Analgesic efficacy | 12 weeks
  Change in Pain score assessed on Numeric Rating Scale (NRS) which ranges from 0 to 10. 0 is no pain and 10 is maximum pain.

SECONDARY OUTCOMES:
Headache days | 12 weeks
  Number of headache days over the course of study period.

CONTACTS AND LOCATIONS:
Overall Officials: Moazzam Ali, Principal Investigator — Pain Medicine Department
Locations (1):
- Pain Medicine Department, Lahore, Pakistan